CLINICAL TRIAL: NCT03023618
Title: Effect Of Stroke Volume Optimization On Complication Rate Of Patients Undergoing Pancreatic Surgery
Brief Title: Fluid Oriented Therapy During Major Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Dr.Andrea Russo, Principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PERILLI-NICE
Record Dates: First submitted 2017-01-01; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Goal Directed Therapy
Keywords: [G09.330.380]

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): patients before 2014, in which fluids were administered without FloTrac monitoring
- case group (Active Comparator): patients after 2014, after management of fluid therapy has been guided by FloTrac parameters as a standard clinical practice (NICE protocol)
  Interventions: Device: FloTrac

INTERVENTIONS:
Device: FloTrac — Stroke Volume has been maintained at 90% of the maximal Stroke Volume as in NICE protocol 2011
  Arms: case group

SUMMARY:
In this "before and after" study we will investigate the potential benefit on postoperative outcomes of a guided fluid therapy with a stroke volume optimization . The NICE protocol has been applied by means of EV1000 monitor and arterial waveform analysis ( Flotrac - Edwards). In the postoperative period overall complications, as well as exitus , will be analyzed and compared with those of a control group underwent the same surgical interventions, with a standard hemodynamic monitoring.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2 patients

Exclusion Criteria:

* Severe Caridiac Disease
* Renal Failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2012-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
complication rate | up to 30 days postoperatively

SECONDARY OUTCOMES:
Duration of hospitalization | an average of 30 days

OTHER OUTCOMES:
amount of intraoperative fluids | an average of 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Valter MD Perilli, PhD, Principal Investigator — Department of Anesthesiology

IPD SHARING:
Plan to Share IPD: Yes